CLINICAL TRIAL: NCT05671237
Title: The Effect of Bilateral Infraorbital+ Infratrochlear Nerve Block on Perioperative Remifentanil Consumption and Postoperative Pain Scores for Rhinoplasty Operations
Brief Title: The Effect of Bilateral Infraorbital+ Infratrochlear Nerve Block for Rhinoplasty Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Reyhan Nil Kırsan, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022/1852
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral infraorbital+infratrochlear block group (Experimental): For this group we will perform bilateral infraorbital+infratrochlear block before surgery
  Interventions: Other: bilateral infraorbital+infratrochlear block
- non-block group (No Intervention): For this group we will start the surgery without performing a block

INTERVENTIONS:
Other: bilateral infraorbital+infratrochlear block — we will perform bilateral infraorbital+infratrochlear nerve block
  Arms: bilateral infraorbital+infratrochlear block group

SUMMARY:
The aim of our study is to examine the effect of bilateral infraorbital and infratrochlear nerve blocks for rhinoplasty operations on perioperative remifentanil need and postoperative pain scores.

DETAILED DESCRIPTION:
Rhinoplasty operations are one of the most applied cosmetic surgeries in the world.

Depending on the procedure type and hemodynamic lability, the quality of the surgical field, perioperative and postoperative complications as well as the success of surgery are affected.To provide improved surgical field quality, controlled hypotension and high concentrations of inhalation anesthetics, magnesium sulfate, remifentanil, clonidine, calcium channel blockers, tranexamic acid, intravenous nitroglycerin have been used.

The American Society of Anesthesiology recommends using regional anesthesia methods and administering multimodal analgesia in every possible surgery. In our study we have performed bilaterral infraorbital an infratrochlear nerve blocks which are main nerves of the nose, for the patients of rhinoplasty. With blocking the infratrochlear and infraorbital nerves we will examine the need for remifentanil during surgery, postoperative pain scores.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing rhinoplasty surgery

Exclusion Criteria:

* Bleeding disorder
* Patient refusal
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Remifentanil consumption | 6 hours
  We will compare the remifentanil consumption for the block performed and non-block group

SECONDARY OUTCOMES:
Surgical bleeding grading | 6 hours
  We will compare the surgical bleeding scores for the block performed and non-block group
Richmond agitation sedation scale | 6 hours
  We will compare the Richmond agitation sedation scale for the block performed and non-block group. +4 Combative +3 Very agitated +2 Agitated +1 Restless 0 Alert and calm -1 Drowsy -2 Light sedation -3 Moderate sedation -4 Deep sedation -5 Unarousable
Numeric rating Scale | 6 hours
  We will compare the numeric rating scale for pain for the block performed and non-block group. The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Post-operative nausea and vomiting | 6 hours
  We will compare the Post-operative nausea and vomiting for the block performed and non-block group
Need for analgesic after surgery | 6 hours
  We will compare the Need for analgesic after surgery for the block performed and non-block group

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boselli E, Bouvet L, Augris-Mathieu C, Begou G, Diot-Junique N, Rahali N, Vertu-Ciolino D, Gerard C, Pivot C, Disant F, Allaouchiche B. Infraorbital and infratrochlear nerve blocks combined with general anaesthesia for outpatient rhinoseptoplasty: A prospective randomised, double-blind, placebo-controlled study. Anaesth Crit Care Pain Med. 2016 Feb;35(1):31-36. doi: 10.1016/j.accpm.2015.09.002. Epub 2015 Nov 5. PMID 26549134
- [Background] Choi H, Jung SH, Hong JM, Joo YH, Kim Y, Hong SH. Effects of Bilateral Infraorbital and Infratrochlear Nerve Block on Emergence Agitation after Septorhinoplasty: A Randomized Controlled Trial. J Clin Med. 2019 May 30;8(6):769. doi: 10.3390/jcm8060769. PMID 31151239
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31151239/